CLINICAL TRIAL: NCT01803191
Title: Randomized Controlled Clinical Trial of Efficacy of Fosfomycin Versus Ciprofloxacin as Antibiotic Prophylaxis Prior to Ultrasound Guided Transrectal Prostate Biopsy
Brief Title: Efficacy Study of Prophylaxis With Fosfomycin Versus Ciprofloxacin Prior Prostate Biopsy
Acronym: BIPROST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: Hospital General Universitario Santa Lucía (Other); Hospital General Universitario Los Arcos del Mar Menor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIPROST; 2012-001031-31 (EudraCT Number)
Record Dates: First submitted 2013-02-14; First posted 2013-03-04 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-03

CONDITIONS: Urinary Tract Infections
Keywords: Transrectal ultrasound-guided prostate biopsy; Bacteriuria; Antibiotic prophylaxis; Prostate-Specific antigen
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria | interventions — Fosfomycin; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fosfomycin 3 g (Experimental): Unique oral dosis of 3 g of fosfomycin 1hour before of biopsy
  Interventions: Drug: Fosfomycin 3 g
- Ciprofloxacin 500 mg (Active Comparator): Unique oral dosis of ciprofloxacin 500 mg before biopsy
  Interventions: Drug: Ciprofloxacin 500 mg

INTERVENTIONS:
Drug: Fosfomycin 3 g — Unique oral dosis of fosfomycin 1 hour before biopsy
  Arms: Fosfomycin 3 g
Drug: Ciprofloxacin 500 mg — Unique oral dosis of ciprofloxacin 500 mg, 1 hour before biopsy
  Arms: Ciprofloxacin 500 mg

SUMMARY:
The purpose of this clinical trial is compare the incidence of symptomatic or asymptomatic bacteriuria after transrectal ultrasound guided prostate biopsy using a single dose of fosfomycin 3 g one hour before the biopsy compared to observed with the use of a single dose of ciprofloxacin 500 mg 1 hour before biopsy.

DETAILED DESCRIPTION:
Transrectal ultrasound guided (TRUS) prostate biopsy is the procedure of choice for the diagnosis of prostate cancer. This technique is usually safe and well tolerated with a low incidence of serious complications. However, one of these complications, the bacterial infection can be complicated and cause urinary sepsis. The investigators have developed different regimens of antibiotic prophylaxis. Most of them include administering oral fluoroquinolones. In this area, approximately 40% of the strains of E. coli are resistant to ciprofloxacin (fluoroquinolone). Therefore, research is warranted alternative prophylactic approaches. Fosfomycin is an antibiotic ancient underused in recent decades that in recent years has been proposed as an alternative treatment for infections caused by multidrug-resistant microorganisms.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with prostate-specific antigen (PSA) values >4 ng/ml or presenting either abnormality in rectal examination
* Patients who accept to participate in the study signing the consent informed form

Exclusion Criteria:

* Allergy to anyone of the study drug
* Intolerance to anyone of the study drug
* Urinary infection with positive uroculture
* Clinical finds suggesting infections
* Antimicrobial treatment during the las 4 weeks
* Patients with vesicle catheter
* Patients in dialysis
* Patients in hemodialysis

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-01-25 (Actual); Study Completion 2016-01-25 (Actual)

PRIMARY OUTCOMES:
Bacteriuria | 28 days
  Positive urine culture(>10000 ufc/ml)

SECONDARY OUTCOMES:
Urinary Tract Infection | 28 days
  clinical symptoms (burning urination, urgent urination, urinary frequency)
Sepsis | 28 days
  Systemic inflammatory response syndrome secondary to urinary tract infection
Pathogens present in urine and antimicrobial resistance | 28 days
Bacteremia | 28 days
  Presence of bacteria in the blood (blood culture positive)
Hematuria | 28 days
  Blood in urine (Complication of transrectal ultrasound guided prostate)
Hemospermia | 28 days
  Blood in the semen (Complication of transrectal ultrasound guided prostate)
Rectal bleeding | 28 days
  Loss of red blood through the anus(Complication of transrectal ultrasound guided prostate)
Urinary retention | 28 days
  Complication of transrectal ultrasound guided prostate
Difficulty for miction | 28 days
  Complication of transrectal ultrasound guided prostate
Genitourinary infections associated to fever (>38ºC) | 28 days
  Fever >38ºC with some of this symptoms: dysuria, polyuria or suprapubic ache
Number of participants with adverse events | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pedro PL Lopez Cubillana, MD, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (3):
- Spain (3):
  - Hospital General Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital General Universitario Los Arcos del Mar Menor, San Javier, Murcia